CLINICAL TRIAL: NCT04740450
Title: Effect of Modified Kinesio Taping Technique on Morbidity After Impacted Third Molar Surgery: Randomized, Placebo-controlled Clinical Trial
Brief Title: Effect of Modified Kinesio Taping Technique on Morbidity After Impacted Third Molar
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Alshaimaa Ahmed shabaan, associate professor in oral & maxillofacial Surgery Department, Fayoum University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KT tape imp
Record Dates: First submitted 2021-02-02; First posted 2021-02-05 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Impacted Third Molar Tooth
Keywords: Impacted third molar; Kinesio taping; swelling

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study side (Experimental): receive KT technique described by Gozluklu et al in 2020
  Interventions: Device: Kinesio taping
- Control side (Placebo Comparator): tapped with wound tape following the same technique
  Interventions: Device: Wound Tape

INTERVENTIONS:
Device: Kinesio taping — skin colored Kinesio-Tex Gold tape, 50 mm _ 5 m (Kinesio Holding Corp, Albuquerque, NM) tapped in technique described by Gozluklu et al in 2020
  Arms: study side
Device: Wound Tape — skin colored wound tape tapped in technique described by Gozluklu et al in 2020
  Arms: Control side

SUMMARY:
Removal of impacted lower third molar is considered as the most common surgical procedure carried out in the oral and maxillofacial Clinics. The surgical removal of the impacted mandibular third molar is usually associated with pain, swelling and inability to open the mouth. Those symptoms reach the maximum intensity between the third to fifth hours postoperatively for the pain and 24 to 48 hours postoperatively for the swelling and then, they gradually diminished until the 7th day postoperatively

DETAILED DESCRIPTION:
Removal of impacted lower third molar is considered as the most common surgical procedure carried out in the oral and maxillofacial Clinics. The surgical removal of the impacted mandibular third molar is usually associated with pain, swelling and inability to open the mouth. Those symptoms reach the maximum intensity between the third to fifth hours postoperatively for the pain and 24 to 48 hours postoperatively for the swelling and then, they gradually diminished until the 7th day postoperatively.

Kinesio taping (KT), also termed ''elastic therapeutic bandage,'' is a popular technique used for the management of postoperative lymphedema after maxillofacial surgery. KT is an elastic therapeutic tape invented by Dr Kase in the 1970s. KT originated from sports medicine and is primarily used to support damaged soft tissues (muscles and joints), helping to reduce pain. KT is considered to regulate the blood and lymph flow and also to remove the congestion of lymphatic fluid or hemorrhage and, thus, has achieved popularity in the control of lymphedema.

Many studies had evaluate the KT technique in reducing the morbidity after surgical removal of third molar. There is a lack of adequate evidence regarding effects of KT techniques versus placebo and the effectiveness of KT with that of other methods and medical agents.

ELIGIBILITY:
Inclusion Criteria:

Age > 18 years, with no systemic disease(s) Bilateral impacted mandibular third molar class II position B on Pell- Gregory classification.

Exclusion Criteria:

* Patients that had any local infection, tobacco use, oral contraceptive, pregnancy, lactation.
* sensitivity to the tapes
* reluctance to shave facial hair (for men)
* known allergies to medication administered in the study,

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2021-06-20 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
postoperative swelling | one week
  Facial swelling was assessed by a three-line measurement method using a flexible plastic tape measure. The corresponding lines were tragus-alanasi (Tr-An; from the most posterior point of the tragus to the most lateral point of the ala nasi), tragus-commissure (Tr-Co; from the most posterior point of the tragus to the most lateral point of the lip commissure), and tragus-pogonion (Tr-Po; from the most posterior point of the tragus to the pogonion) distances. These measurements were performed with the patient sitting at 90° straight position with physiologic rest position of the mandible.

SECONDARY OUTCOMES:
pain | one week
  VAS measure
Preoperative and postoperative mouth opening | one week
  measurement of the maximal distance between the cutting edge of the right maxillary and right mandibular central incisors with a caliper.

CONTACTS AND LOCATIONS:
Overall Officials: Alshaimaa a Mohamed, phd, Principal Investigator — Fayoum University
Locations (1):
- Faculty of Dentistry, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gozluklu O, Ulu M, Gozluklu HO, Yilmaz N. Comparison of Different Kinesio Taping Techniques After Third Molar Surgery. J Oral Maxillofac Surg. 2020 May;78(5):695-704. doi: 10.1016/j.joms.2019.12.026. Epub 2020 Jan 7. PMID 32008990
- [Background] Jaron A, Jedlinski M, Grzywacz E, Mazur M, Trybek G. Kinesiology Taping as an Innovative Measure against Post-Operative Complications after Third Molar Extraction-Systematic Review. J Clin Med. 2020 Dec 9;9(12):3988. doi: 10.3390/jcm9123988. PMID 33317073
- [Background] Tatli U, Benlidayi IC, Salimov F, Guzel R. Effectiveness of kinesio taping on postoperative morbidity after impacted mandibular third molar surgery: a prospective, randomized, placebo-controlled clinical study. J Appl Oral Sci. 2020;28:e20200159. doi: 10.1590/1678-7757-2020-0159. Epub 2020 Jul 13. PMID 32667383